CLINICAL TRIAL: NCT00484575
Title: Inhaled Sevoflurane Compared to Intravenous Sedation Post Coronary Artery Bypass Grafting
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Peter Sackey, MD, PhD, Dept of Physiology and Pharmacology, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-000293-23
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2007-06

CONDITIONS: Myocardial Reperfusion Injury; Atrial Fibrillation
Keywords: Sevoflurane; CABG; cardioprotection; AnaConDa
MeSH Terms: conditions — Myocardial Reperfusion Injury; Atrial Fibrillation | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol (Active Comparator): propofol for sedation minimum 2 hours in CTICU after CABG
  Interventions: Drug: propofol
- sevoflurane (Experimental): Sevoflurane via AnaConDa for minimum 2 hours in CTICU after CABG
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — given by infusion via AnaConDa for sedation with target MAAS 2-3
  Other Names: Sevorane
  Arms: sevoflurane
Drug: propofol — propofol given intravenously for sedation in control group
  Arms: propofol

SUMMARY:
Inhaled sevoflurane during coronary artery bypass grafting (CABG) reduces postoperative Troponin levels and may be associated with improved outcome. A dose-response effect has been demonstrated by de Hert et al, with greatest reductions of Troponin when Sevoflurane was used during the entire operation, as compared to Sevoflurane during parts of the operation.

Sevoflurane, as other inhaled anesthetic agents, is sedative in low doses. Postoperative sedation after CABG is currently achieved with intravenous propofol.

A new simplified method of administration of isoflurane or sevoflurane has been developed and tested by members of the research group. The Anesthetic Conserving Device is a modified heat-moisture exchanger (HME) that permits direct infusion of sevoflurane to the airway, where it is vaporized in an evaporator rod in the device.

The primary aim (and primary hypothesis)of the current trial is to examine if postoperative sedation with sevoflurane after CABG is associated with improved cardiac outcome, measured as reduced levels of Troponin, BNP and reduced incidence of cardiac events, such as atrial fibrillation, need for inotropic drugs and myocardial infarction, compared with conventional propofol sedation.

Other end-points of the trial are potential renal (protective) effects measured with cystatin C levels, need for dialysis but also measurements of inorganic fluorides in serum, as well as environmental aspects of sevoflurane sedation in a Cardiothoracic Intensive Care Unit. Furthermore, potential differences in ICU memories and well-being during stay in the intensive Care Unit will be investigated via patient questionnaires.

Besides routine blood sampling, plasma will be saved for later analysis of inflammatory mediators (biobank).

DETAILED DESCRIPTION:
Sevoflurane, an inhaled anesthetic is currently recommended for anesthesia during coronary artery bypass grafting (CABG).

Inhaled sevoflurane during CABG reduces postoperative Troponin levels and may be associated with improved outcome. A dose-response effect of Sevoflurane cardioprotection has been demonstrated by de Hert et al, with greatest reductions of Troponin when Sevoflurane was used during the entire operation, as compared to Sevoflurane during parts of the operation or not at all.

Postoperative sedation after CABG is currently achieved with intravenous propofol.

Sevoflurane, as other inhaled anesthetic agents, is sedative in low doses. A new simplified method of administration of isoflurane or sevoflurane has been developed and tested by members of the research group. The Anesthetic Conserving Device (AnaConDa®) is a modified heat-moisture exchanger (HME) that permits direct infusion of sevoflurane to the airway, where it is vaporized in an evaporator rod in the device. Studies of isoflurane sedation with the AnaConDa® have shown good sedation effects and short wake-up times.

The primary aim (and primary hypothesis)of the current trial is to examine if postoperative sedation with sevoflurane after CABG is associated with improved cardiac outcome, measured as reduced levels of Troponin, BNP and reduced incidence of cardiac events, such as atrial fibrillation, need for inotropic drugs and myocardial infarction, compared with conventional propofol sedation.

Other end-points of the trial are potential renal (protective) effects measured with cystatin C levels, need for dialysis but also measurements of inorganic fluorides in serum, as well as environmental aspects of sevoflurane sedation in a Cardiothoracic Intensive Care Unit. Furthermore, potential differences in ICU memories and well-being during stay in the intensive Care Unit will be investigated via patient questionnaires.

Besides routine blood sampling, plasma will be saved for later analysis of inflammatory mediators (biobank).

Methods:

120 patients planned for CABG (without valve surgery) will be enrolled in the trial. Patients with malignant hyperthermia are excluded, as well as patients with need for mechanical circulation support.

Routine anesthesia and CABG will be followed by randomisation to either inhaled sevoflurane or intravenous propofol. Patients will be transferred from the operating room to the Cardiothoracic Intensive Care Unit (CICU)with propofol sedation. Upon arrival to the CICU sedation will according to randomisation will replace propofol.

Thereafter patients will be kept sedated according to the MAAS Scale until vital parameters are stable and extubation criteria are fulfilled or for a maximum of 48 hours. Time from arrival at CICU to extubation, as well as time from termination of sedative to extubation will be measured. Total time in CICU will be recorded as well as time from arrival to discharge criteria are fulfilled.

Troponin, BNP, Creatinine, Cystatin C, CRP will be measured before CABG, and at regular time intervals postoperatively. A blood sample for storage of plasma will be taken 12 hours postoperatively, preliminary for measurement of interleukin activity as this may be attenuated by inhaled anesthetics. Hemodynamics will be recorded during CICU care, as well as need for inotropic drugs, cardioversion, arrythmias or adverse events.

Environment will be monitored with dosimeter measurements and with spectrophotometry.

After extubation patients will be monitored regarding cognitive recovery during the first hour. When discharged from the CICU, patients will receive a questionnaire in order to describe the memory panorama from the ICU stay after 1-2 days.

ELIGIBILITY:
Inclusion Criteria:

* Planned coronary artery bypass grafting

Exclusion Criteria:

* Combined heart valve surgery
* Malignant Hyperthermia
* Postoperative need for mechanical circulation support

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Troponin levels | 2 days

SECONDARY OUTCOMES:
renal function | 1 week
ambient sevoflurane levels | 2 days
cognitive function/memory panorama post ICU | 1 week
attenuation of inflammatory response | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Sackey, MD, PhD, Principal Investigator — Karolinska Institutet, Institution of Physiology and Pharmacology, Section for Anesthesia and Intensive Care Medicine; Jan-Olof Hellström, MD, Principal Investigator — Karolinska Institutet, Institution of Physiology and Phrmacology, Section for Anesthesia and Intensive Care; Anders Öwall, MD, PhD, Principal Investigator — Karolinska University Solna, Department of Cardiothoracic Anesthesia and Intensive Care
Locations (1):
- Karolinska University Hospital Solna, Cardiothoracic Intensive Care Unit, Stockholm, Sweden